CLINICAL TRIAL: NCT03715504
Title: A Phase I, First-in-human, Open-label, Dose Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Oral TP-3654 in Patients With Advanced Solid Tumors
Brief Title: Study of TP-3654 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-3654-101
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumors
Keywords: Sumitomo Dainippon Pharma Oncology SDPO; Solid Tumor; Advanced Malignancy; First in Human; Phase 1; Cancer
MeSH Terms: conditions — Neoplasms | interventions — TP 3654

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm TP-3654 (Experimental): TP-3654 by oral administration
  Interventions: Drug: TP-3654

INTERVENTIONS:
Drug: TP-3654 — oral PIM inhibitor

SUMMARY:
TP-3654 is an oral PIM inhibitor. This is a Phase 1, open-label, dose-escalation, safety, pharmacokinetics, and pharmacodynamic study, with a purpose of determining the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of oral TP-3654 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of oral TP-3654 in patients with advanced solid tumors.

Secondary Objectives:

* To establish the pharmacokinetic (PK) profile of orally administered TP-3654
* To observe patients for any evidence of antitumor activity of TP-3654 by objective radiographic assessment
* To study the pharmacodynamic effects of TP-3654 therapy
* To establish the Recommended Phase 2 Dose (RP2D) for future studies with TP-3654

ELIGIBILITY:
Inclusion Criteria:

* 1. Have a histologically confirmed diagnosis of advanced metastatic, progressive or unresectable solid tumor

  2. Be refractory to, or intolerant of, established therapy known to provide clinical benefit for their condition.

  3. Have 1 or more tumors measurable or evaluable as outlined by modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

  4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2

  5. Have a life expectancy greater than or equal to 3 months

  6. Be greater than or equal to 18 years of age

  7. Have a negative pregnancy test (if female of childbearing potential) and not currently nursing

  8. Have acceptable liver function:

  a. Bilirubin less than or equal to 1.5x upper limit of normal (ULN) (unless associated with Gilbert's syndrome b. Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) and alkaline phosphatase less than or equal to 2.5x upper limit of normal (ULN) *If liver metastases are present, then less than or equal to 5x ULN is allowed.

  9. Have acceptable renal function:

  a. Calculated creatinine clearance greater than or equal to 30 mL/min

  10. Have acceptable hematologic status:

  a. Absolute Neutrophil Count (ANC) greater than or equal to 1500 x10^9/L b. Platelet count greater than or equal to 100,000 x 10^9/L c. Hemoglobin greater than or equal to 8 g/dL

  11. Have acceptable coagulation status:
  1. Prothrombin time (PT) within 1.5 x normal limits
  2. Activated partial thromboplastin time (aPTT) within 1.5 x normal limits

     12. Be nonfertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use an effective method of contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation and for 3 months (males) and 6 months (females) after the last study drug dose. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

     13. Have read and signed the Institutional Review Board (IRB)-approved informed consent form prior to any study related procedure. (In the event that the patient is re-screened for study participation or a protocol amendment alters the care of an ongoing patient, a new informed consent form must be signed.)

     Exclusion Criteria:
* 1. History of congestive heart failure (CHF), Cardiac disease, myocardial infarction within the past 6 months prior to Cycle 1 Day 1, left ventricular ejection fraction <45% by echocardiogram, unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG) within 14 days prior to Cycle 1 Day 1

  2. Have a corrected QT interval (using Fridericia's correction formula) (QTcF) of >450 msec in men and >470 msec in women

  3. Presence of symptomatic central nervous system metastatic disease or disease that requires local therapy such as radiotherapy, surgery, or increasing dose of steroids within the prior 2 weeks.

  4. Have severe chronic obstructive pulmonary disease with hypoxemia (defined as resting 02 saturation of less than or equal to 90% breathing room air). The use of supplemental oxygen with nasal cannula to reach >90% saturation will not preclude study participation.

  5. Have undergone major surgery, other than diagnostic surgery, within 2 weeks prior to Cycle 1 Day 1

  6. Have active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy

  7. Received treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within 28 days or 5 half-lives, whichever occurs first, prior to study entry (6 weeks for nitrosoureas or Mitomycin C)

  8, Are unwilling or unable to comply with procedures required in this protocol

  9. Have known infection with human immunodeficiency virus, hepatitis B, or hepatitis C. Patients with history of chronic hepatitis that is currently not active are eligible.

  10. Have a serious nonmalignant disease (eg, hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor

  11. Are currently receiving any other investigational agent

  12. Have exhibited allergic reactions to a similar structural compound, biological agent, or formulation

  13. Have a medical conditional such as Crohn's disease or have undergone significant surgery to the gastrointestinal tract that could impair absorption or that could result in short bowel syndrome with diarrhea due to malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) and treatment emergent adverse events | 28 days
Determine maximum tolerated dose (MTD) | 20 months
  MTD will be determined based upon toxicity grades which are defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Recommended Phase 2 Dose of TP-3654 | 23 months
  To establish the Recommended Phase 2 Dose (RP2D) for future studies with TP-3654, MTD data to be reviewed
Determine antitumor activity of TP-3654 | 20 months
  Assess for tumor burden by radiological assessment (computed tomography [CT] imaging) using RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sumitomo Dainippon Pharma Oncology, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (3):
- United States (3):
  - MD Anderson, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia